CLINICAL TRIAL: NCT00146211
Title: A Multicenter, Double Blind, Randomized, Parallel Group, Placebo-Controlled Trial of Ethyl-EPA (Miraxion™) in Subjects With Mild to Moderate Huntington's Disease
Brief Title: TREND-HD - A Trial of Ethyl-EPA (Miraxion™) in Treating Mild to Moderate Huntington's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amarin Neuroscience Ltd (Industry)
Collaborators: Huntington Study Group (Network)
Responsible Party: Ira Shoulson, MD/Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN01.01.0011
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Huntington Disease
Keywords: Trial; ethyl-EPA; Miraxion™; treating; mild; moderate; Huntington's
MeSH Terms: conditions — Huntington Disease; Lymphoma, Follicular | interventions — eicosapentaenoic acid ethyl ester; Docosahexaenoic Acids

INTERVENTIONS:
Drug: Ethyl-EPA (Miraxion™)

SUMMARY:
This study is designed to determine the effect of 2 gram/day of ethyl-EPA on motor (movement) signs and symptoms of Huntington disease.

DETAILED DESCRIPTION:
Multi-center, double blind, placebo-controlled study with parallel groups of outpatients with early, symptomatic Huntington's disease. Participants will be randomized to receive 1 gram twice daily (2 gram/day total daily dose) of active study drug or placebo. The 6-month placebo-controlled phased will be followed by a subsequent 6-month open-label extension phase with all subjects receiving 1 gram twice daily (2 grams/day total daily dose) of active study drug.

ELIGIBILITY:
Inclusion Criteria:

* Clinical features of Huntington's disease (HD) and confirmatory family history of HD, and/or CAG repeat expansion greater than or equal to 36
* Ambulatory, not requiring skilled nursing care (total functional capacity [TFC] greater than or equal to 7)
* Chorea score of at least 2 in one extremity (UHDRS)
* Maximal dystonia less than or equal to 2 and maximal bradykinesia less than or equal to 2
* 35 years of age or older of either gender
* Must be on stable dosages of non-competitive NMDA receptor antagonists, and/or antiepileptic medications for 60 days prior to baseline
* Females of child-bearing potential must use adequate birth control

Exclusion Criteria:

* History of established diagnosis of tardive dyskinesia
* Clinical evidence of unstable medical or psychiatric illness
* Clinically significant active and unstable psychotic disease (hallucinations or delusions)
* Major depression (Beck Depression Inventory [BDI]-II Score greater than 20) at Screening Visit
* Suicidal ideation (BDI-II item 9 greater than or equal to 2) at Screening Visit
* History of clinically significant substance abuse within 12 months of Baseline Visit
* Pregnant/lactating women
* Participation in other drug studies within 60 days prior to Baseline Visit
* Previous participation in any investigational study of ethyl-EPA (Miraxion™)
* Use of aspirin at daily dosage greater than 325 mg/day
* Exclusionary Drugs (within 6 months Baseline Visit): Depot neuroleptics
* Exclusionary Drugs (within 60 days Baseline Visit): Omega-3 supplementation, tetrabenazine or reserpine, high dose and/or variable dose oral anti-psychotic medications, steroid (other than topical), selenium supplements greater than 55 mcg/day, lithium, benzodiazepines (except for low dose), anticoagulants

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2005-09; Primary Completion 2007-08 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To compare with placebo the effect of ethyl-EPA on the Total Motor Score-4 component (TMS) of the Unified Huntington's Disease Rating Scale (UHDRS) over a 6-month period of observation.

SECONDARY OUTCOMES:
To compare with placebo the effect of ethyl-EPA over a 6-month period of observation on, 1) Chorea (UHDRS Total Motor Score Scale); 2) Total Motor Score component (TMS) of the UHDRS; and, 3) Clinical Global Impression (CGI) score.

CONTACTS AND LOCATIONS:
Overall Officials: Ira Shoulson, MD, Principal Investigator — Huntington Study Group/University of Rochester; Christopher Ross, MD, PhD, Principal Investigator — Huntington Study Group/Johns Hopkins University School of Medicine; Blair Leavitt, MD, Principal Investigator — Huntington Study Group/University of British Columbia
Locations (41):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Institute of Neurodegenerative Disorders, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Kansas City, Kansas
  - Hereditary Neurological Disease Centre, Wichita, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University, Boston, Massachusetts
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Albany Medical College, Albany, New York
  - North Shore-LIJ Health System, Manhasset, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Ohio State University Parkinson's Center, Columbus, Ohio
  - Penn State Milton & Hershey Medical College, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee-Memphis, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Glenrose Rehab Hospital, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of British Columbia, London, Ontario
  - The Centre for Addiction and Mental Health, Markham, Ontario
  - Hotel-Dieu Hospital-CHUM, Montreal, Quebec

REFERENCES:
- [Derived] Huntington Study Group TREND-HD Investigators. Randomized controlled trial of ethyl-eicosapentaenoic acid in Huntington disease: the TREND-HD study. Arch Neurol. 2008 Dec;65(12):1582-9. doi: 10.1001/archneur.65.12.1582. PMID 19064745
- See also: Related Info — http://www.Huntington-Study-Group.org